CLINICAL TRIAL: NCT05074121
Title: N-acetylcysteine for Attenuation of COVID Symptomatology
Brief Title: NAC for Attenuation of COVID-19 Symptomatology
Acronym: NACinCOVID2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge Health Alliance (Other)
Collaborators: The Thoracic Foundation (Unknown); Alturix (Unknown)
Responsible Party: Principal Investigator, Melisa Lai-Becker, Chief, CHA Everett Emergency Department; Director, CHA Division of Medical Toxicology, Cambridge Health Alliance
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Record Dates: First submitted 2021-10-05; First posted 2021-10-12 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Lower Respiratory Infection; SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere; Oxidative Stress
Keywords: acetylcysteine; N-acetylcysteine; N-acetyl-cysteine; NAC; glutathione
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blinded Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and study team members will be masked to whether a participant is receiving the study drug or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC (Experimental): Group receiving intervention/study drug NAC
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Group receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine
  Other Names: NAC; N-acetyl-cysteine; Acetylcysteine
  Arms: NAC
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether oral NAC is effective at attenuating COVID-19 disease symptom severity and duration of symptoms.

DETAILED DESCRIPTION:
STUDY DESIGN: Randomized double-blinded placebo-controlled trial

ELIGIBILITY

Inclusion criteria:

* age 18 years and older
* participants will need daily access to use of a smartphone for at least six weeks from time of enrollment
* Positive COVID-19 test within 10 days of date of enrollment
* not already hospitalized for treatment of COVID

Exclusion criteria:

* pregnant
* already hospitalized for treatment of COVID

PROTOCOL

* 50:50 randomization: half of participants will take NAC, half will take placebo
* Participants will take NAC/placebo following this outpatient protocol:
* 2400 mg x 1 PO then
* 1200 mg PO BID x 14 days
* Participants will complete an online symptom-tracker for six weeks (daily for three weeks, weekly for three weeks)

ELIGIBILITY:
Inclusion Criteria:

* positive COVID test <= 7 days of enrollment

Exclusion Criteria:

* pregnant
* already hospitalized due to COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Symptom severity | 24 weeks starting the day after enrollment
  Severity of symptoms
Symptom duration | 24 weeks starting the day after enrollment
  Length in days of symptoms

SECONDARY OUTCOMES:
Need for higher level of care/hospitalization | 24 weeks starting the day after enrollment
  Comparison between groups of rates of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge Health Alliance, Everett, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data used for publication
Supporting Information: Study Protocol, ICF
Time Frame: Available six months after publication for one year
URL: http://www.NACinCOVID.info